CLINICAL TRIAL: NCT02138344
Title: Assessment of Neuropathic Pain
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: EK-04/2006 / PB_2016-02051
Record Dates: First submitted 2014-05-12; First posted 2014-05-14 (Estimated); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Spinal Cord Injury + Peripheral Nerve Diseases
MeSH Terms: conditions — Spinal Cord Injuries; Peripheral Nervous System Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | US Export: No

GROUPS / COHORTS (3):
- SCI subjects: Chronic and traumatic SCI subjects
- Healthy control subjects
- Subjects with peripheral nerve diseases

SUMMARY:
Development of neuropathic pain is one of the most disabling sequels after spinal cord injury (SCI) and in peripheral nerve diseases. The functionality of the pain pathway in humans as well as its plastic changes following SCI can be assessed in vivo by surface electrophysiological recordings and functional magnetic resonance imaging after noxious heat stimulation of the skin. Aims: a) establishing a clinically applicable assessment of the pain pathway and characterizing its changes as a consequence of SCI and in peripheral nerve diseases in an objective manner, b) characterizing plastic changes in the pain pathway in SCI patients with neuropathic pain and in patients with peripheral nerve diseases and relating them to the development of neuropathic pain syndromes.

ELIGIBILITY:
Inclusion Criteria:

* Uninjured
* Scord injured subjects
* Subjects with peripheral nerve diseases
* Patients resident in Switzerland

Exclusion Criteria:

* Presence of any central psychiatric disorder (that precludes subject from giving informed and voluntary consent)
* For fMRI measurements: "yes" for any item in the MR-risk questionnaire
* Patients resident outside from Switzerland

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with SCI and peripheral nerve diseases
Sampling Method: Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2006-04-01 (Actual); Primary Completion 2024-09-27 (Actual); Study Completion 2024-09-27 (Actual)

PRIMARY OUTCOMES:
Pain, sensory and autonomic assessments | 2 - 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Curt, Armin, MD, Zurich, Canton of Zurich, Switzerland